CLINICAL TRIAL: NCT00570141
Title: Case Study Documentation of Subjects With Either Diabetic Foot Ulcers or Venous Stasis Ulcers Being Treated With OASIS
Brief Title: OASIS Wound Matrix (Oasis) Mechanism of Action
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Innes Cargill, PhD, Director, Clinical Affairs Tissue Management, Healthpoint, Ltd.
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 9310-002-004
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Results first posted 2010-08-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Foot Ulcers (DFU); Venous Stasis Ulcers (VSU)
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OASIS Wound Matrix (Oasis) (Active Comparator): This is a single arm study with only the test article Oasis used on all subjects
  Interventions: Device: OASIS Wound Matrix

INTERVENTIONS:
Device: OASIS Wound Matrix — OASIS (an acellular biomaterial that supports tissue repair with a scaffold-like matrix having a natural structure and composition).

SUMMARY:
OASIS Wound Matrix (Oasis) will be applied to wounds, with sequential biopsy of healing wounds to explore the mechanism of action.

DETAILED DESCRIPTION:
Wound types will be Diabetic Foot Ulcers (DFU) and Venous Stasis Ulcers (VSU).

ELIGIBILITY:
Inclusion Criteria:

* Diabetic foot ulcer (DFU) or venous stasis ulcer (VSU) of the leg, with certain restrictions on size, duration and underlying health

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the study medications or their components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Payne, M.D., Principal Investigator — Bay Pines VA Healthcare System; Carl Van Gils, DPM, CWS, Principal Investigator — Dixie Regional Medical Center Wound Clinic; Davin Haraway, DO, Principal Investigator — Sparks Regional Medical Center
Locations (3):
- United States (3):
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Bay Pines VA Healthcare System, St Louis, Missouri
  - Dixie Regional Medical Center Wound Clinic, St. George, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- OASIS Wound Matrix (Oasis): All subjects in this study were treated with Oasis®, there were no other test articles used in this study.
Period: Overall Study
Arm/Group | OASIS Wound Matrix (Oasis)
Started | 13
Completed | 10
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Missed visits | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | OASIS Wound Matrix (Oasis)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 63.5 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13
Wound Type [Number; unit: Participants]
  DFU | 7
  VSU | 6

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Wound Area From Baseline After 12 Weeks of Treatment or Until Wound Closure, Whichever Occurred First.
Description: Wound measurements were made weekly, spaced 7 +/- 1 day apart, up to 12 weeks or until the wound healed, whichever occurred first.
  The final measurement taken was subtracted from the baseline to assess the decrease in wound area after treatment.
  Final calculation is mean baseline measurement minus final measurement at 12 weeks (or when wound healed, whichever occurred first)
Time Frame: Baseline and weekly up to 12 weeks
Population: Analysis was Per Protocol
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | OASIS Wound Matrix (Oasis)
Number analyzed (Participants) | 13
cm2
  Diabetic Foot Ulcers (DFU) | 1.3 (0.6)
  Venous Stasis Ulcers (VSU) | 3.6 (2.2)

2. Primary Outcome: Percent Wounds Closed
Description: Wound healing was assessed weekly, spaced 7 +/- 1 day apart, up to 12 weeks or until the wound healed, whichever occurred first.
  The outcome value was based on the percent of wounds which were closed at the end of the study (at 12 weeks). The percent wounds closed were calculated for each wound type: Diabetic Foot Ulcers (DFU) and Venous Stasis Ulcers (VSU).
Time Frame: baseline and 12 weeks
Population: Analysis was Per Protocol
Measure: Number; unit: Percent of Wounds Closed
Arm/Group | OASIS Wound Matrix (Oasis)
Number analyzed (Participants) | 13
Percent of Wounds Closed
  Diabetic Foot Ulcers (DFU) | 50.0
  Venous Stasis Ulcers (VSU) | 66.7

ADVERSE EVENTS:
Arm/Group | OASIS Wound Matrix (Oasis)
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OASIS Wound Matrix (Oasis) (N=13)
Follicular swelling (Infections and infestations) | 1 (1) — Infected insect bite - not related to test article
Urinary Tract Infection (Infections and infestations) | 1 (1) — not related to test article
Infection left foot 1st metatarsal head (Infections and infestations) | 1 (1) — Injury - not related to test article
Osteomyelitis left foot 1st metatarsal head (Infections and infestations) | 1 (1) — Osteomyelitis - not related to test article
Cellulitis left foot ulcer (Infections and infestations) | 1 (1) — Cellulitis of the foot, non-test ulcer - not related to the test article
Open wound (Injury, poisoning and procedural complications) | 1 (1) — Head wound - not related to test article
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) — Biopsy pain - not related to test article
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — Right leg pain - not related to test article
Blister 2nd toe, left foot, with loose nail (Skin and subcutaneous tissue disorders) | 1 (1) — Blister - not related to test article
Achilles tendon repair (Surgical and medical procedures) | 1 (1) — Tendon operation - not related to test article
Ulcer - right foot 5th toe medially (Vascular disorders) | 1 (1) — Skin ulcer - non-target ulcer - not related to test article

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No